CLINICAL TRIAL: NCT03134417
Title: Parathyroid Hormone and Cardiometabolic Outcomes in Obesity: Role of Magnesium and Vitamin D Supplementation
Brief Title: Magnesium and Vitamin D Supplementation and Cardiometabolic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1407002973
Record Dates: First submitted 2017-04-07; First posted 2017-05-01 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Overweight and Obesity; Vitamin D Deficiency; Magnesium Deficiency; Cardiovascular Risk Factor
MeSH Terms: conditions — Overweight; Obesity; Vitamin D Deficiency; Magnesium Deficiency | interventions — Vitamin D; Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin D and magnesium (Experimental): Daily oral vitamin D (1000 IU) and magnesium (360 mg) supplement
  Interventions: Dietary Supplement: Vitamin D and magnesium
- Vitamin D (Active Comparator): Daily oral vitamin D (1000 IU) supplement
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Daily oral placebo (cellulose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D and magnesium — Daily vitamin D and magnesium supplements are given to participants daily for 12 weeks.
  Arms: Vitamin D and magnesium
Dietary Supplement: Vitamin D — Daily vitamin D supplements are given to participants daily for 12 weeks.
  Arms: Vitamin D
Dietary Supplement: Placebo — Daily placebo are given to participants daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of a combined vitamin D and magnesium supplementation on parathyroid hormone and cardiometabolic health in persons living with obesity.

DETAILED DESCRIPTION:
Individuals living with obesity are at a higher risk of cardiometabolic abnormalities and high circulating parathyroid hormone. There is evidence suggesting that vitamin D may play a role in cardiovascular health outcomes; however, the research is currently inconclusive. Magnesium is a cofactor of vitamin D metabolism, and the prevalence of concurrent vitamin D and magnesium deficiency is high. This study aims to investigate the effect of vitamin D and magnesium supplements in individuals who are overweight and obese on parathyroid hormone and cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* BMI range 25-40 kg/m2
* 30-70 years of age

Exclusion Criteria:

* Presence of any acute illness in the past month
* Pre-existing chronic medical conditions or medications know to influence energy, vitamin D, magnesium and calcium metabolism, levels of blood glucose, lipids and blood pressure
* Individuals taking vitamin D and magnesium supplement greater than the Recommended Daily allowance
* Participants taking any medications or have disease known to influence calcium or bone metabolism

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Serum parathyroid hormone | 12 weeks

SECONDARY OUTCOMES:
Inflammatory cytokines | 12 weeks
Lipid profile | 12 weeks
Blood pressure | 12 weeks
Serum osteocalcin | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University Nutrition Sciences Research Lab, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dall RD, Cheung MM, Shewokis PA, Altasan A, Volpe SL, Amori R, Singh H, Sukumar D. Combined vitamin D and magnesium supplementation does not influence markers of bone turnover or glycemic control: A randomized controlled clinical trial. Nutr Res. 2023 Feb;110:33-43. doi: 10.1016/j.nutres.2022.12.005. Epub 2022 Dec 22. PMID 36640582